CLINICAL TRIAL: NCT03214991
Title: Circulating Tumor DNA as a Prognostic Marker in Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ji Kon Ryu (Other)
Responsible Party: Sponsor-Investigator, Ji Kon Ryu, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: 1704-108-847
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood circulating tumor DNA in patients with pancreatic cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the usefulness of circulating tumor DNA as a prognostic factor in patients with pancreatic cancer.

DETAILED DESCRIPTION:
There is currently no strong prognostic factor in pancreatic cancer. K-ras is the most commonly mutated gene in pancreatic cancer, with a mutation rate of 75% to 95%. These high mutation rates are expected to be useful for diagnosis and prognostic factors in future. Currently, K-ras mutation tests are often performed in tissues, and there are various limitations, in particular, limited obtaining of sufficient tissues. In this regard, analyzing the prognosis of pancreatic cancer through non-invasive blood testing has significant advantages. And Prognosis analysis through blood tests can be done through blood circulating tumor DNA. The relationship between prognosis and blood circulating tumor DNA has already been studied in other cancers such as colorectal cancer, and there have been several studies in pancreatic cancer. However, there are not many research results yet, and there are cases in which the results differ from study to study. Therefore, the purpose of this study is to compare the overall survival of patients with pancreatic cancer diagnosed by EUS-FNA according to the presence and amount of blood circulating tumor DNA with K-ras mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer through EUS-FNA.

Exclusion Criteria:

* Severe mental illness
* Severe co-morbidity (ESRD, Advanced COPD, severe Heart failure, poorly controlled blood sugar)
* Pregnancy
* Patients who have received chemotherapy
* Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pancreatic cancer through EUS-FNA.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 48 months
  Comparison of overall survival rates between patients with and without blood-circulating tumor DNA

SECONDARY OUTCOMES:
Overall survival rate according to the amount of blood circulating tumor DNA | 48mo
  Overall survival rate according to the amount of blood circulating tumor DNA
K-ras mutation | 48 months
  The concordance rate of K-ras mutation in EUS-FNA specimen and K-ras mutation in blood circulating tumor DNA
Overall survival rate (EUS-FNA) | 48 months
  Overall survival rate with or without K-ras mutation of EUS-FNA specimen
Overall survival rate (K-ras mutation type, circulating tumor DNA) | 48 months
  Overall survival rate according to K-ras mutation type in blood circulating tumor DNA
Overall survival rate (K-ras mutation type, EUS-FNA) | 48 months
  Overall survival rate according to K-ras mutation type in EUS-FNA specimen

CONTACTS AND LOCATIONS:
Overall Officials: Ji Kon Ryu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No